CLINICAL TRIAL: NCT05250687
Title: MR Guided Focused Ultrasound Versus Radiotherapy for Palliative Pain Treatment in Patients With Bone Metastases
Brief Title: MR Guided Focused Ultrasound vs Radiotherapy for Palliative Pain Tx in Bone Metastases
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insigthec is no longer seeking support of the device used for this clinical trial
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-62458
Record Dates: First submitted 2022-02-01; First posted 2022-02-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Bone Metastases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- MR guided high intensity focused ultrasound (MR-HIFU) (Experimental): MRHIFU treatment will be delivered using the ExAblate 2100 System (INSIGHTEC, Tirat Carmel, Israel), which is an FDA-approved device for pain palliation of bone metastases.
  Interventions: Procedure: MR- High intensity focused ultrasound
- External beam radiation therapy (EBRT) (Active Comparator): Patients will undergo radiotherapy for painful bone metastases.
  Interventions: Radiation: External beam radiotherapy

INTERVENTIONS:
Procedure: MR- High intensity focused ultrasound — The intervention treatment is MR-HIFU, which will be given as a standalone treatment. MRHIFU treatment will be delivered using the ExAblate 2100 System (INSIGHTEC, Tirat Carmel, Israel), which is an FDA-approved device for pain palliation of bone metastasesThe ExAblate focused ultrasound device operates in conjunction with an MRI machine. Gadavist is being administered intraveneously as contrast medium for MRI.
  Other Names: MR-HIFU
  Arms: MR guided high intensity focused ultrasound (MR-HIFU)
Radiation: External beam radiotherapy — Standard of care for pain palliation of bone metastases consists of single fraction external beam radiotherapy of 8-16 Gray (Gy) or a multi-fraction regime of 20 Gy in 5 fractions, 24 Gy in 6 fractions or 30 Gy in 10 fractions. The radiation schedule is at the discretion of the treating radiation oncologist.
  Other Names: EBRT
  Arms: External beam radiation therapy (EBRT)

SUMMARY:
This is a prospective, single-center, randomized study directly comparing outcomes after MR guided high intensity focused ultrasound (MR HIFU) or external beam radiation therapy (EBRT) treatment of painful bone metastases.

DETAILED DESCRIPTION:
The primary purpose of this study is to see if MR guided high intensity focused ultrasound (MR-HIFU) treats bone pain faster than the standard radiation therapy (External beam radiation therapy: EBRT) and to evaluate the patient's pain experience 14 days after completion of the treatment. The secondary purpose is to evaluate the outcomes of the pain, side effects, and quality of life and survival in the first 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Painful metastatic bone lesions, with NRS > 4 documented at screening visit
3. Pain from target lesion is distinguishable from other lesions*
4. Target lesion lovation is accessible for MR-HIFU and EBRT**
5. Target lesion is visible om MR or CT imaging obtained < 3 months prior to screening, with a maximum diameter of 8 cm.
6. Reasonable performance score (KPS > 50% or ECOG <3)
7. Life expectancy > 3 months as determined by the study PI or referring oncologist
8. Ability to understand and the willingness to personally sign the written IRB-approved informed consent document

   * Solitary painful metastatic bone lesion or multiple metastatic lesions with one predominantly painful target lesion (≥2 points higher pain score than other lesions).

     * e.g.: Extremities, pelvis (os pubis, os ilium, os ischium, sacrum, acetabulum), shoulders, in selected cases ribs and sternum

Exclusion Criteria:

1. Previous surgery, radiation, HIFU, or other local therapy on the target location
2. Neurological symptoms due to nerve involvement of target lesion
3. Need for surgery of targeted location due to (impending) pathological fracture
4. Unavoidable critical structures or dense tissues in target area*
5. Curative intention of treatment plan
6. Patients with contraindication for MR imaging such as implanted metallic devices that are not MRI - safe, size limitations, claustrophobia, etc.
7. Patients with known intolerance or allergy to MR contrast agent (gadolinium chelates) including advanced kidney disease (GFR <30mL/min/1.73 m^2) or on dialysis
8. Pregnant and nursing patients will be excluded from the study because of a contraindication to administering MRI contrast agents to these patients
9. Patients unable to receive general anesthesia, as determinded by anesthesiologist, study PI or referring oncologist
10. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (can be up to 4 hrs of total table time) via self report
11. Participant enrolled in another clinical interventional study related to bone metastases treatment or pain relief treatment
12. Clinically relevant medical history or physical findings that could interfere with the patient's safety as judged by the treating physician

    * as judged by the operator. e.g.: nerve bundles, skin, extensive scarring, non-targeted bones, air (e.g. hollow viscera), (external) fixation device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants that achieve a complete response (CR) or partial response (PR) | 14 days after treatment
  Complete response (CR): Complete response is defined as a pain score of zero at the treated site with no concomitant increase in analgesic intake (stable or reducing analgesics in daily oral morphine equivalents). Partial Response (PR): Partial response is to be defined as any of the following: Pain reduction of 2 or more points at the treated site on a 0-10 scale without analgesic increase; or analgesic dose reduction of 25% or more in daily morphine equivalent from baseline without an increase in pain.

SECONDARY OUTCOMES:
Patient-reported pain scores - Pain Diary | 1 month
  Patient reported pain scores will be based on a Numeric Rating Scale (NRS) (from 0 to 10) 0 = no pain and 10= worst pain. Assessed using the patient pain diary from treatment day to 1 month after completion treatment.
Patient-reported pain scores - BPI (Brief Pain Inventory) | on baseline, at 2 and 4 weeks, and at 3 and 6 months
  The BPI measures pain interference on seven 0-10 integer subscales, as well as the mean of the seven subscales.
Physician-reported adverse events | on baseline, at 2 and 4 weeks, and at 3 and 6 months
  Assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0; we will report the number of pathologic fractures at the site of treatment
Patient-reported quality of life - EORTC QLQ-BM22 | on baseline, at 2 and 4 weeks, and at 3 and 6 months
  During follow up, patient will received quality of life questionnaire on baseline, at 2 and 4 weeks, and at 3 and 6 months after completion of treatment.
Patient-reported quality of life - EORTC QLQ-C15-PAL | on baseline, at 2 and 4 weeks, and at 3 and 6 months
  During follow up, patient will received quality of life questionnaire on baseline, at 2 and 4 weeks, and at 3 and 6 months after completion of treatment.
Patient-reported quality of life - EQ-5D-5L | on baseline, at 2 and 4 weeks, and at 3 and 6 months
  During follow up, patient will received quality of life questionnaire on baseline, at 2 and 4 weeks, and at 3 and 6 months after completion of treatment.
Patient-reported quality of life - PGIC | on baseline, at 2 and 4 weeks, and at 3 and 6 months
  During follow up, patient will received quality of life questionnaire on baseline, at 2 and 4 weeks, and at 3 and 6 months after completion of treatment. Patient Global Impression of Change scale has a single question with a 7 point likert scale about overall improvement after treatment assessing change in pain, from "Much Better" to "Much Worse"
Local tumor control | 3 and 6 months after completion of treatment
  Assessed using CT and/or MRI imaging at three and/or six months after completion of treatment
Anxiety and depression scores | on baseline, at 2 and 4 weeks, and at 3 and 6 months
  Assessed by the Hospital Anxiety and Depression Scale (HADS). This measures anxiety and depression separately on seven four-point (0-3) subscales, giving total scores from 0-21 for both constructs.

CONTACTS AND LOCATIONS:
Overall Officials: Pejman Ghanouni, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No